CLINICAL TRIAL: NCT02352129
Title: Prognostic Value of Myocardial Fibrosis Quantified Using CMR in Patient With Dilated Cardiomyopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-A00887-34
Record Dates: First submitted 2015-01-21; First posted 2015-02-02 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Cardiomyopathy, Dilated
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardiomyopathy dilated patient (Experimental): Cardiomyopathy dilated patients wil be evalueted by CMR using T1 mapping technique to evalueted the level myocardial fibrosis
  Interventions: Other: CMR using T1 mapping technique
- healthy subjects (Active Comparator): healthy subject wil be evaluated by CMR using T1 mapping technique to know the baseline of myocardial fibrosis in healthy subjects
  Interventions: Other: CMR using T1 mapping technique

INTERVENTIONS:
Other: CMR using T1 mapping technique — the level of myocardial fibrosis for patient suffering of cardiomyopathy dilated will be quantified using CMR T1 mapping technique

SUMMARY:
: Fibrosis, in general, is a scarring process, which is characterized by fibroblast accumulation and excess deposition of extracellular matrix (ECM) proteins, which leads to distorted organ architecture and function. The contribution of fibrogenesis to impaired cardiac function is increasingly recognized. The fibrotic ECM causes increased stiffness and induces pathological signaling within cardiomyocytes resulting in progressive cardiac failure. Also, the excessive ECM impairs mechano-electric coupling of cardiomyocytes and increases the risk of arrhythmias. But today patient treatment and prognosis is based on ejection fraction quantification, QRS duration, and symptoms.

Hypothesis: the increased level of fibrosis quantified using T1 mapping technique, compared with normal value, is of prognostic value in patient with dilated cardiomyopathies under optimal treatment.

Methods: 330 patients are planned to be included and followed for 2 years

ELIGIBILITY:
Inclusion Criteria:

* patient with dilated cardiomyopathy and typical symptoms of cardiac insufficiency at the time of the diagnosis: oedemas of lower limbs, dyspnoea, asthenia.
* and of a reduction in the fraction of ventricular ejection left (awkward) 45 % measured in echocardiography ( modified Simpson biplane) and associated with a volume télédiastolic volume superior to the normal in echocardiography: > 90ml / m2 ( modified Simpson biplane).

Exclusion Criteria:

* Patients to whom the dysfunction VG is secondary or in a secondary overload of pressures in a HTA or a severe valvulopathie is in a coronary infringement(achievement), proved by histories of infarct or gestures(movements) of revascularisation (bypass(decking), stent) and or coronary hurts at least bi tronculaires significant the severity of which can explain the ventriculaire failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Prognostic value of the increased level of myocardial fibrosis | two years
  The long-term forecast of the patients affected by CMD will be estimated by the survival without event. The events considered in this study are included in an associating combined criterion:
  * Death(Deaths), whatever is its cause.
  * The heart transplant
  * Hospitalization for cardiac cause, including acute(sharp) cardiac insufficiency, disorder(confusion) of the rhythm, required by rehabilitation of the treatment(processing), the thrombus ventriculaire left, cerebrovascular accident.
  * Palpitation ventriculaire steady (ventriculaire extrasystole > 120 pulsation for minutes more than 30 on Holter of 24 hours(12 pm)).
  * Palpitation ventriculaire not steady

SECONDARY OUTCOMES:
hemodynamic consequences of the increased level of myocardial fibrosis | txw years
  The quantity of interstitial fibrosis at the time of the diagnosis will be correlated to the indicators of the reshaping left ventriculaire measured in echocardiography: decrease of more than 10 % of the fraction of ejection over 2 years or increase of the volume télédiastolique furthermore of 20ml / the year.

CONTACTS AND LOCATIONS:
Overall Officials: alexis JACQUIER, MD, Principal Investigator — Assistance Public Hôpitaux de marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Cadour F, Quemeneur M, Biere L, Donal E, Bentatou Z, Eicher JC, Roubille F, Lalande A, Giorgi R, Rapacchi S, Cortaredona S, Tradi F, Bartoli A, Willoteaux S, Delahaye F, Biene SM, Mangin L, Ferrier N, Dacher JN, Bauer F, Leurent G, Lentz PA, Kovacsik H, Croisille P, Thuny F, Bernard M, Guye M, Furber A, Habib G, Jacquier A. Prognostic value of cardiovascular magnetic resonance T1 mapping and extracellular volume fraction in nonischemic dilated cardiomyopathy. J Cardiovasc Magn Reson. 2023 Feb 6;25(1):7. doi: 10.1186/s12968-023-00919-y. PMID 36747201